CLINICAL TRIAL: NCT06240273
Title: Assessment of Therapeutic Potential of Stigma Maydis (Cornsilk) on Metabolic Syndrome
Acronym: cornsilk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Silk syndrome
Record Dates: First submitted 2024-01-17; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Hypertension; Obesity; Insulin Resistance; Diabetes; Cornsilk powder; Dyslipidemia
MeSH Terms: conditions — Metabolic Syndrome; Hypertension; Obesity; Insulin Resistance; Diabetes Mellitus; Dyslipidemias

STUDY DESIGN:
Intervention Model Description: Single group Assignment Case-control Study
Masking Description: None (open-label) Participants Groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metabolic Syndrome patients (Experimental): Cornsilk (Stigma maydis) is used for preventing symptoms of metabolic syndrome patients Dietary Intervention: Cornsilk Extract Dosage: 2g/day
  Interventions: Dietary Supplement: Corn silk powder

INTERVENTIONS:
Dietary Supplement: Corn silk powder — Corn silk (CS) is abundant in phenolic compounds, especially flavonoids. It also contains proteins, vitamins, carbohydrates, calcium, potassium, magnesium, sodium salts, volatile oils, sterols like sitosterol and stigmasterol, alkaloids, and saponins. Numerous studies have explored the pharmacological activities associated with CS.
  Other Names: stigma maydis

SUMMARY:
Over the past two decades, there has been an increase in the number of people with nutrition related maladies due to changes in their dietary habits and lifestyle. Cardiovascular disease, type 2 diabetes, metabolic syndrome, obesity, and cancer have emerged as prominent contributors to both illness and death, particularly as the population continues to age. The mortality figures for cardiovascular disease and diabetes varied between 179.8 to 765.2 per 100,000 individuals, with the most elevated rates observed in poor nations. The occurrence of metabolic syndrome was markedly prevalent, spanning from 19% to 45%. The incidence of overweight and obesity (defined by a body mass index ≥25 kg/m2) has surged to concerning levels across many countries in the region, ranging from 25% to 82%, with a higher occurrence among women. Due to side effects of allopathic treatments and increase in nutrition knowledge people are more inclined to natural therapies. Subsequently, corn silk with nutraceutical properties may provide an effective alternative therapy to alleviate symptoms and decrease healthcare loss. Cornsilk, the often-overlooked byproduct of maize cultivation, is rich in bioactive compounds, including flavonoids, polysaccharides, and vitamins, cornsilk has shown promising effects in promoting health and wellness.

DETAILED DESCRIPTION:
Background:

Over the past two decades, there has been an increase in the number of people with nutrition related maladies due to changes in their dietary habits and lifestyle. Cardiovascular disease, type 2 diabetes, metabolic syndrome, obesity, and cancer have emerged as prominent contributors to both illness and death, particularly as the population continues to age. The mortality figures for cardiovascular disease and diabetes varied between 179.8 to 765.2 per 100,000 individuals, with the most elevated rates observed in poor nations. The occurrence of metabolic syndrome was markedly prevalent, spanning from 19% to 45%. The incidence of overweight and obesity (defined by a body mass index ≥25 kg/m2) has surged to concerning levels across many countries in the region, ranging from 25% to 82%, with a higher occurrence among women. Due to side effects of allopathic treatments and increase in nutrition knowledge people are more inclined to natural therapies. Subsequently, corn silk with nutraceutical properties may provide an effective alternative therapy to alleviate symptoms and decrease healthcare loss. Cornsilk, the often-overlooked byproduct of maize cultivation, is rich in bioactive compounds, including flavonoids, polysaccharides, and vitamins, cornsilk has shown promising effects in promoting health and wellness.

Hypothesis: Stigma maydis (corn silk) has a potential to manage metabolic syndrome.

Objective: To assess the therapeutic effect of Stigma maydis (corn silk) against metabolic syndrome.

Methodology: Cornsilk powder will be procured from a local market. The proximate analysis and total phenolic content of the product will be performed and then capsules of powder will be prepared to be consumed by the participants. A total of 40 subjects (20 in treatment group and 20 in control group) will be selected and capsules will be added to their diets (1000mg twice a day). After a trial of 45 days, the patients will be assessed. Assessment will include anthropometric measurements, blood pressure, lipid profile analysis and blood sugar levels which will be monitored before and after the trial and finally, the data collected will be analyzed by using SPSS 25 by paired sample t test. P value ≤ 0.05 will be considered significant.

Expected outcomes: Stigma maydis (corn silk) capsules will prove to have therapeutic potential against obesity, hypertension, glucose intolerance and dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Waist Circumference of ≥40 inches in males and ≥35 inches for females
* Subjects having fasting total cholesterol level of ≥ 200 mg/dl or LDL cholesterol ≥ 130 mg/dl.
* Fasting Blood Glucose ≥110mg/dl.
* SBP ≥ 130/ ≥ 85 mmHg

Exclusion Criteria:

* Participants aged 55 or above • Participants who have less than two risk factors

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-20 (Estimated); Primary Completion 2024-04-20 (Estimated); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
Lipid profile will be assessed before and after the trial. | 45 days
  The change in lipid profile, after 45 days intervention of corn silk extract, will be assessed. The value will be closed to optimized values.
waist circumference will be measured before and after the trial. | 45 days
  the change in weight will be measured after 45 days of corn silk extract intervention. The value will be close to normal ranges.
Blood pressure will be assessed before and after the trial. | 45 days
  The change in systolic and diastolic blood pressure will be measured after 45 days intervention of corn silk extract. The values will become close to optimized levels.
Fasting glucose level will be assessed before and after the trial. | 45 days
  The change in fasting glucose levels will be assessed after 45 days intervention of corn silk extract powder. The values will be become close to optimized levels

CONTACTS AND LOCATIONS:
Overall Officials: Dr. M. Asif Ali, PhD, Principal Investigator — University of Veterinary and Animal Sciences, lahore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shahzad MK, Amir Shahzad M, Qadeer U, Mehmood A. Investigation of phytochemical profiling and therapeutic effects of corn silk against diabetes in human male subjects. Pak J Pharm Sci. 2022 Nov;35(6(Special)):1699-1703. PMID 36861231
- [Background] Shi S, Yu B, Li W, Shan J, Ma T. Corn silk decoction for blood lipid in patients with angina pectoris: A systematic review and meta-analysis. Phytother Res. 2019 Nov;33(11):2862-2869. doi: 10.1002/ptr.6474. Epub 2019 Aug 18. PMID 31423665